CLINICAL TRIAL: NCT04383938
Title: Study of APR-246 in Combination With Pembrolizumab in Subjects With Solid Tumor Malignancies
Brief Title: Phase 1/2 Study of APR-246 in Combination With Pembrolizumab in Subjects With Solid Tumor Malignancies
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Aprea Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: A20-11195
Record Dates: First submitted 2020-05-07; First posted 2020-05-12 (Actual); Results first posted 2025-05-13 (Actual); Last update posted 2025-05-13 (Actual); Status verified 2025-05

CONDITIONS: Bladder Cancer; Gastric Cancer; Non Small Cell Lung Cancer; NSCLC; Urothelial Carcinoma; Advanced Solid Tumor
Keywords: Pembrolizumab; APR-246; Aprea; eprenetapopt
MeSH Terms: conditions — Urinary Bladder Neoplasms; Stomach Neoplasms; Carcinoma, Non-Small-Cell Lung; Carcinoma, Transitional Cell | interventions — eprenetapopt; pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Safety Lead In-Phase 1 Dose Level 1 (Experimental): APR-246 4.5g/d with pembrolizumab 200 mg IV (day 3) every 21 days in patients with advanced non-CNS primary tumors
  Interventions: Drug: APR-246 (eprenetapopt) + Pembrolizumab
- Expansion 1- Gastric Cancer (Experimental): APR-246 4.5 g/d (days 1-4) with pembrolizumab 200 mg IV (day 3) every 21 days in patients with advanced gastric or GEJ tumors
  Interventions: Drug: APR-246 (eprenetapopt) + Pembrolizumab
- Expansion 2- Bladder Cancer (Experimental): APR-246 4.5 g/d (days 1-4) with pembrolizumab 200 mg IV (day 3) every 21 days in patients with advanced bladder or urothelial tumors
  Interventions: Drug: APR-246 (eprenetapopt) + Pembrolizumab
- Expansion 3 -NSCLC (Experimental): APR-246 4.5 g/d (days 1-4) with pembrolizumab 200 mg IV (day 3) every 21 days in patients with advanced NSCLC.
  Interventions: Drug: APR-246 (eprenetapopt) + Pembrolizumab

INTERVENTIONS:
Drug: APR-246 (eprenetapopt) + Pembrolizumab — APR-246 D1-4 + Pembrolizumab D3

SUMMARY:
A phase 1/2, open-label, study to determine the safety and preliminary efficacy of APR-246 in combination with pembrolizumab in subjects with solid tumor malignancies. The study will include a safety lead-in portion followed by a phase 2 expansion portion in specific disease groups.

DETAILED DESCRIPTION:
This is a phase 1/2, open-label, study to determine the safety and preliminary efficacy of APR-246 (eprenetapopt) in combination with pembrolizumab in subjects with solid tumor malignancies. In the safety lead-in part of study (phase 1), the safety and the recommended phase 2 dose (RP2D) of APR-246 will be investigated.

In the expansion part of the study (phase 2), both safety and efficacy for the combination therapy will be investigated in the 3 cohorts.

ELIGIBILITY:
Inclusion Criteria:

1. Signed informed consent form (ICF) and ability to comply with protocol requirements.
2. Known tumor TP53 mutation status from recent or archival sample.
3. Histologically and/or cytologically confirmed solid tumor malignancy

   1. Safety lead in- Advanced non-central nervous system (CNS) primary tumors that have progressed after first line treatment, who are intolerant to first line treatment, or who are unable to receive first line treatment, and for whom pembrolizumab, or pembrolizumab-based therapy is considered appropriate
   2. Expansion 1- Patients with a confirmed diagnosis of advanced gastric or gastroesophageal junction (GEJ) tumors that have progressed after first line treatment, who are intolerant to first line treatment, or who are unable to receive first line treatment
   3. Expansion 2- Patients with a confirmed diagnosis of advanced bladder/urothelial tumors that have progressed after first line treatment, or who are intolerant to first line treatment, or who are unable to receive first line treatment with cisplatin-based chemotherapy.
   4. Expansion 3- Confirmed diagnosis of advanced non-small cell lung cancer (NSCLC) previously treated with anti-PD-1 or anti-PD-L1 therapy.
4. Adequate organ function

   1. Creatinine clearance > 30 mL/min
   2. Total serum bilirubin < 1.5 × upper limit of normal (ULN) unless due to Gilbert's syndrome, tumor involvement, hemolysis or considered an effect of regular blood transfusions
   3. Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) < 3 × ULN, unless due to involvement by the underlying malignancy.
5. Projected life expectancy of ≥ 12 weeks.
6. Age ≥ 18 years at the time of signing the ICF.
7. Eastern Cooperative Oncology Group (ECOG) performance status of 0, 1 or 2
8. In the expansion portion, measurable disease meeting the following criteria:

   1. At least 1 lesion of ≥10 mm in the longest diameter (LD) for a non-lymph node or ≥15 mm in the short-axis diameter for a lymph node that is serially measurable according to RECIST 1.1.
   2. Lesions that have had external beam radiotherapy or loco-regional therapies such as radiofrequency ablation must show subsequent evidence of substantial size increase (ex. 20% increase in LD) to be deemed a target lesion.
9. Negative serum or urine pregnancy test prior to study treatment initiation in female subjects of childbearing potential.
10. Women of childbearing potential and men with female partners of childbearing potential must be willing to use an effective form of contraception

Exclusion Criteria:

1. Known history of untreated human immunodeficiency virus (HIV)/HIV with a detectable viral load or active hepatitis B or active hepatitis C infection.
2. Cardiac abnormalities
3. Concomitant malignancies or previous malignancies with less than a 1-year disease-free interval at the time of signing consent.
4. Pregnancy or lactation.
5. Active uncontrolled systemic infection.
6. An autoimmune condition requiring ≥ 10 mg (or equivalent corticosteroid) prednisone daily, or any other systemic immunosuppressive treatment within 28 days of first dose of study therapy.
7. Known history of active tuberculosis.
8. Current (non-infectious) pneumonitis, or a history of pneumonitis that required steroids.
9. A live vaccine administered within 30 days of the first dose of study treatment.
10. Receipt of any investigational product within 14 days or 5 half-lives prior to study treatment initiation, whichever is shortest.
11. Prior intolerance to pembrolizumab or other anti-PD-1/PD-L1 agents.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2020-06-25 (Actual); Primary Completion 2022-04-30 (Actual); Study Completion 2022-04-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joachim Gullbo, MD, Study Director — Theradex Oncology
Locations (8):
- United States (8):
  - Mayo Clinic, Phoenix, Arizona
  - Mayo Clinic, Jacksonville, Florida
  - Massachusetts General Hospital, Boston, Massachusetts
  - Dana Farber Cancer Center, Boston, Massachusetts
  - Mayo Clinic, Rochester, Minnesota
  - Washington University, St Louis, Missouri
  - Vanderbilt University, Nashville, Tennessee
  - MD Anderson Cancer Center, Houston, Texas

REFERENCES:
- [Derived] Park H, Shapiro GI, Gao X, Mahipal A, Starr J, Furqan M, Singh P, Ahrorov A, Gandhi L, Ghosh A, Hickman D, Gallacher PD, Wennborg A, Attar EC, Awad MM, Das S, Dumbrava EE. Phase Ib study of eprenetapopt (APR-246) in combination with pembrolizumab in patients with advanced or metastatic solid tumors. ESMO Open. 2022 Oct;7(5):100573. doi: 10.1016/j.esmoop.2022.100573. Epub 2022 Sep 7. PMID 36084396

RESULTS

PARTICIPANT FLOW:
Groups:
- Experimental: Safety Lead In: Patients with advanced solid tumors. APR 4.5 g/day intravenously (IV) on days 1-4 with pembrolizumab 200 mg IV on day 3 in each 21-day cycle
- Experimental: Expansion 1: Patients with advanced gastric cancer. APR 4.5 g/day intravenously (IV) on days 1-4 with pembrolizumab 200 mg IV on day 3 in each 21-day cycle
- Experimental: Expansion 2: Patients with advanced urothelial/bladder cancer. APR 4.5 g/day intravenously (IV) on days 1-4 with pembrolizumab 200 mg IV on day 3 in each 21-day cycle
- Experimental: Expansion 3: Patients with advanced NSCLC. APR 4.5 g/day intravenously (IV) on days 1-4 with pembrolizumab 200 mg IV on day 3 in each 21-day cycle
Period: Overall Study
Arm/Group | Experimental: Safety Lead In | Experimental: Expansion 1 | Experimental: Expansion 2 | Experimental: Expansion 3
Started | 6 | 8 | 5 | 21
Completed | 6 | 6 | 5 | 20
Not Completed | 0 | 2 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Baseline characteristics are presented by cohort.
Groups:
- Experimental: Expansion 1 Patients With Advanced Gastric Cancer.: Patients with advanced gastric cancer. APR 4.5 g/day intravenously (IV) on days 1-4 with pembrolizumab 200 mg IV on day 3 in each 21-day cycle
- Experimental: Expansion 3 Patients With Advanced NSCLC: Patients with advanced NSCLC. APR 4.5 g/day intravenously (IV) on days 1-4 with pembrolizumab 200 mg IV on day 3 in each 21-day cycle
- Total: Total of all reporting groups
Arm/Group | Experimental: Safety Lead In | Experimental: Expansion 1 Patients With Advanced Gastric Cancer. | Experimental: Expansion 2 | Experimental: Expansion 3 Patients With Advanced NSCLC | Total
Number analyzed (Participants) | 6 | 8 | 5 | 21 | 40
Age, Continuous [Median (Full Range); unit: years] | 58 [35 to 85] | 67 [27 to 79] | 67 [55 to 75] | 67 [54 to 85] | 66 [27 to 85]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 1 | 1 | 13 | 17
  Male | 4 | 7 | 4 | 8 | 23
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 1 | 0 | 1 | 1 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 4 | 4
  White | 5 | 7 | 3 | 16 | 31
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 1 | 0 | 2
Region of Enrollment [Number; unit: participants]
  United States | 6 | 8 | 5 | 21 | 40

OUTCOME MEASURES:

1. Primary Outcome: To Evaluate the Safety of APR-246 in Combination With Pembrolizumab in Subjects With Solid Tumors.
Description: To determine the Frequency of treatment-emergent adverse events (TEAEs), and serious adverse events (SAEs) related to APR-246 in combination with pembrolizumab.
Time Frame: Through study completion, approximately 1 year
Population: Data is presented by cohort/arm. 3 out of the 40 overall patients did not receive treatment on study. 37 total patients were analyzed
Measure: Number; unit: participants
Arm/Group | Experimental: Safety Lead In | Experimental: Expansion 1 | Experimental: Expansion 2 | Experimental: Expansion 3
Number analyzed (Participants) | 6 | 6 | 5 | 20
participants | 6 | 6 | 5 | 20

2. Primary Outcome: To Confirm the Recommended Phase 2 Dose (RP2D) for APR-246 in Combination With Pembrolizumab
Description: To determine the dose of APR-246 to be selected for the expansion phase based on the occurence of dose limiting toxicities (DLTs) experienced during the safety assessment period
Time Frame: Through safety lead in period, during cycle 1 (approximately 21 days)
Population: Experimental: Safety Lead In" Arm/Group was analyzed for this Outcome Measure
Measure: Number; unit: g/d
Arm/Group | Experimental: Safety Lead In
Number analyzed (Participants) | 6
g/d | 4.5

ADVERSE EVENTS:
Time Frame: 13 months
Description: Data is presented by overall study enrollment and not by cohort.
Arm/Group | Experimental: Safety Lead In | Experimental: Expansion 1 | Experimental: Expansion 2 | Experimental: Expansion 3
All-Cause Mortality (participants affected / at risk) | 5/6 | 4/6 | 2/5 | 10/20
Serious Adverse Events (participants affected / at risk) | 1/6 | 4/6 | 3/5 | 7/20
Other Adverse Events (participants affected / at risk) | 6/6 | 5/6 | 5/5 | 20/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Experimental: Safety Lead In (N=6) | Experimental: Expansion 1 (N=6) | Experimental: Expansion 2 (N=5) | Experimental: Expansion 3 (N=20)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 3
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 2
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Disease Progression (General disorders) | 1 | 1 | 0 | 0
Pain (General disorders) | 0 | 1 | 1 | 0
Asthenia (General disorders) | 0 | 0 | 0 | 1
Pyrexia (General disorders) | 0 | 0 | 0 | 1
Abdominal Pain (Gastrointestinal disorders) | 1 | 0 | 1 | 0
Abdominal pain lower (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Abdominal Pain upper (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Hypotension (Vascular disorders) | 0 | 0 | 1 | 1
Embolism (Vascular disorders) | 0 | 1 | 0 | 0
Blood bilirubin Increased (Investigations) | 0 | 0 | 0 | 1
Blood Creatinine increased (Investigations) | 0 | 0 | 0 | 1
Acute Kidney Injury (Renal and urinary disorders) | 0 | 1 | 0 | 0
Haematuria (Renal and urinary disorders) | 0 | 0 | 0 | 1
Anemia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0
Atrial Fibraltion (Cardiac disorders) | 0 | 0 | 0 | 1
Hyperbilirubinemia (Hepatobiliary disorders) | 0 | 1 | 0 | 0
Urinary tract Infection (Infections and infestations) | 0 | 0 | 0 | 1
Hypernatraemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Dizziness (Nervous system disorders) | 1 | 0 | 0 | 0
Confusional State (Psychiatric disorders) | 0 | 0 | 0 | 1
Pelvic Pain (Reproductive system and breast disorders) | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Experimental: Safety Lead In (N=6) | Experimental: Expansion 1 (N=6) | Experimental: Expansion 2 (N=5) | Experimental: Expansion 3 (N=20)
Nasuea (Gastrointestinal disorders) | 3 | 2 | 4 | 6
Vomiting (Gastrointestinal disorders) | 1 | 1 | 4 | 6
Constipation (Gastrointestinal disorders) | 1 | 1 | 3 | 5
Abdominal Pain (Gastrointestinal disorders) | 4 | 0 | 3 | 1
Proctalgia (Gastrointestinal disorders) | 0 | 0 | 2 | 0
Retching (Gastrointestinal disorders) | 0 | 2 | 0 | 0
Stomatitis (Gastrointestinal disorders) | 0 | 2 | 0 | 0
Diarrhea (Gastrointestinal disorders) | 0 | 2 | 3 | 2
Dizziness (Nervous system disorders) | 1 | 1 | 4 | 9
Tremor (Nervous system disorders) | 1 | 1 | 1 | 2
Headache (Nervous system disorders) | 0 | 0 | 2 | 2
Neuropathy peripheral (Nervous system disorders) | 0 | 1 | 1 | 0
Paraesthesia (Nervous system disorders) | 0 | 0 | 0 | 2
Somnolence (Nervous system disorders) | 0 | 2 | 0 | 0
Decreased Appetite (Metabolism and nutrition disorders) | 2 | 3 | 1 | 6
Hyponatremia (Nervous system disorders) | 0 | 1 | 2 | 3
Hyperglycemia (Nervous system disorders) | 0 | 0 | 1 | 3
Dehydration (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 2 | 1
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 0 | 2 | 0
Malnutrition (Metabolism and nutrition disorders) | 0 | 0 | 2 | 0
Fatigue (General disorders) | 4 | 1 | 4 | 3
Pyrexia (General disorders) | 0 | 0 | 2 | 2
Asthenia (General disorders) | 0 | 0 | 1 | 1
Chills (General disorders) | 0 | 0 | 2 | 0
Disease progression (General disorders) | 1 | 1 | 0 | 0
Oedema Peripheral (General disorders) | 1 | 0 | 0 | 1
Pain (General disorders) | 0 | 1 | 1 | 0
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 6
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 0
Pulmonary Embolisim (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 2
Alanine aminotransferase increased (Investigations) | 1 | 2 | 1 | 2
Aspartate aminotransferase increased (Investigations) | 0 | 1 | 1 | 3
Blood alkaline phosphatase increased (Investigations) | 4 | 0 | 1 | 2
Blood creatinine increased (Investigations) | 1 | 1 | 0 | 1
Blood thyroid stimulating hormone increased (Investigations) | 0 | 1 | 0 | 1
Lymphocyte count decreased (Investigations) | 0 | 0 | 1 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 0 | 1 | 0
Muscular Weakness (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 3
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 3 | 1
Anaemia (Blood and lymphatic system disorders) | 1 | 1 | 4 | 3
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 2
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 2
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 1
Hypotension (Vascular disorders) | 0 | 1 | 1 | 2
Hypertension (Vascular disorders) | 1 | 0 | 0 | 1
Confusional state (Psychiatric disorders) | 0 | 0 | 0 | 3
Anxiety (Psychiatric disorders) | 0 | 0 | 1 | 1
Insomnia (Psychiatric disorders) | 0 | 1 | 1 | 1
Urinary tract infection (Infections and infestations) | 0 | 0 | 1 | 3
Atrial Fibrillation (Cardiac disorders) | 0 | 0 | 0 | 2
Sinus Tachycardia (Cardiac disorders) | 0 | 0 | 2 | 0
Acute Kidney Injury (Renal and urinary disorders) | 0 | 1 | 1 | 0
Vision Blurred (Eye disorders) | 0 | 0 | 0 | 2
Vertigo (Ear and labyrinth disorders) | 1 | 0 | 0 | 1
Abdominal Pain Upper (Gastrointestinal disorders) | 1 | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-03-13): https://cdn.clinicaltrials.gov/large-docs/38/NCT04383938/Prot_SAP_000.pdf